CLINICAL TRIAL: NCT03061461
Title: A Prospective, Randomized, Double-blind, Placebo Controlled, Parallel Group, Single Center Trial to Assess the Efficacy and Safety of Radial Extracorporeal Shock Wave Therapy in Subjects With Chronic Soft Tissue Wounds
Brief Title: Radial Extracorporeal Shock Wave Therapy for Chronic Soft Tissue Wounds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kuala Lumpur General Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Harikrishna K.Ragavan Nair, Head, Wound Care Unit, Dept. of Internal Medicine, KualaLGH, Kuala Lumpur General Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NMRR-16-1660-32178 (IIR)
Record Dates: First submitted 2017-02-19; First posted 2017-02-23 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Wound of Skin
Keywords: Extracorporeal shock wave therapy; ESWT; Radial extracorporeal shock wave therapy; rESWT; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT), no blinding of therapists applying the treatments, blinding of patients, blinding of evaluators.
  Partial cross-over design: patients in the control group will be offered to be treated with rESWT starting three months after the last sham treatment. This will guarantee that every patient will receive a real rESWT treatment independent of blind allocation to one of the treatment groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A medical assistant in the Wound Care Unit, Dept on Internal Medicine, Kuala Lumpur Hospital (Kuala Lumpur, Malaysia) will allocate interventions by means of opaque sealed envelopes that will be marked according to the allocation schedule. The medical assistant will be unaware of the size of the blocks.
  The randomized intervention assignment as outlined above will be concealed from both patients and health care staff until recruitment will be complete and irrevocable.
  Therapists applying the treatments will not be blinded.
  All assessments before the first treatment (baseline) and during the follow-up period (either three months after start of the treatments or until complete epithelialization, respectively) will be performed by assessors blind to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- rESWT (Active Comparator): Treatment of chronic wounds with the Swiss DolorClast (Electro Medical Systems S.A., Nyon, Switzerland) and the EvoBlue handpiece as follows:
  * Use of the 15-mm applicator or the 36-mm applicator of the Swiss DolorClast according to the individual wound size.
  * Six treatment sessions, two treatment sessions per week.
  * 1000 radial shock waves per cm^2 wound and treatment session.
  * Energy flux density 0.07 mJ/mm^2 (i.e., setting of the air pressure of the Swiss DolorClast at 2 bar when using the 15-mm applicator, and at 4 bar when using the 36-mm applicator).
  * Frequency of the radial shock waves set at 15 Hz.
  Interventions: Device: rESWT
- Sham rESWT (Sham Comparator): Treatment of chronic wounds with the Swiss DolorClast (Electro Medical Systems S.A., Nyon, Switzerland) and the placebo EvoBlue handpiece of the Swiss DolorClast (that looks and sounds like the EvoBlue handpiece of the Swiss DolorClast, but does not generate radial shock waves) as follows:
  * Use of the 15-mm applicator or the 36-mm applicator of the Swiss DolorClast according to the individual wound size.
  * Six treatment sessions, two treatment sessions per week.
  * 1000 sham radial shock waves per cm^2 wound and treatment session.
  * Energy flux density 0.00 mJ/mm^2 (setting of the air pressure of the Swiss DolorClast at 2 bar when using the 15-mm applicator, and at 4 bar when using the 36-mm applicator).
  * Frequency of the sham radial shock waves set at 15 Hz.
  Interventions: Device: Sham rESWT

INTERVENTIONS:
Device: rESWT — All patients will receive standard care as follows:
  1. Wounds will be cleaned with distilled water and applied with collagen gel or collagen sheet on the wound and then closed with foam/gauze or gamgee.
  2. The clean wounds will be assessed using the TIME concept.
  3. Treatment with rESWT.
  4. Subsequently the wounds will be cleansed with distilled water, and collagen and glycerine gel will be applied and covered with adhesive dressings (Melolin, Smith & Nephew, Inc. Advanced Wound Management; Fort Worth, TX, USA).
  In addition, patients in arm "rESWT" will receive rESWT between Steps 2 and 3 of standard care as outlined in arm description "rESWT".
  Arms: rESWT
Device: Sham rESWT — All patients will receive standard care as follows:
  1. Wounds will be cleaned with distilled water and applied with collagen gel or collagen sheet on the wound and then closed with foam/gauze or gamgee.
  2. The clean wounds will be assessed using the TIME concept.
  3. Treatment with sham rESWT.
  4. Subsequently the wounds will be cleansed with distilled water, and collagen and glycerine gel will be applied and covered with adhesive dressings (Melolin).
  In addition, patients in arm "Sham rESWT" will receive sham rESWT between Steps 2 and 3 of standard care as outlined in arm description "Sham rESWT".
  Arms: Sham rESWT

SUMMARY:
This study tests the hypothesis that radial extracorporeal shock wave therapy (rESWT) as performed by Zoech (JATROS Orthop 2009;(1):46-47) is effective and safe in treatment of chronic soft tissue wounds, and is statistically significantly more effective than sham-treatment of chronic soft tissue wounds.

DETAILED DESCRIPTION:
Zoech (2009) treated in a feasibility study a total of n=18 patients affected by 21 ulcers in Stage IA or IIA (according to Armstrong and colleagues, Diabetes Care 1998;21:855-859) with repetitive radial extracorporeal shock wave therapy (rESWT) using the Swiss DolorClast device (Electro Medical Systems S.A., Nyon, Switzerland). The wounds had been observed for more than 6 weeks. In nine cases the wounds were located in non-loaded areas such as the edge of the foot, or appeared after previous toe amputation. In 12 cases the wounds were located on the sole, the toes or the heel; in these cases the average area of the wounds was 351 mm^2 (116 to 599 mm^2). Local wound treatment consisted of regular debridement by scalpel, followed by disinfection with sterile saline solution and application of wet treatment adequate to the stage of the wounds. Depending on the amount of secretion, the depth of the ulcer and the healing stages, different bandage materials were used. Besides this, rESWT was applied at intervals depending on the size and the depth of the ulcers, once or twice a week for three to six weeks, with 1,000 impulses per cm^2 and treatment session with positive energy flux density (EFD) of 0.1 mJ/mm^2. To this end ulcers were covered with sterile drape in order to avoid direct contact of ultrasound jelly and the handpiece of the rESWT device with the ulcers. After further disinfection with sterile saline solution, bandage was applied. The state of the ulcers was documented photographically at regular intervals and the size of the ulcers were evaluated with digital image analysis. Wounds were evaluated after the first, second and third week. Zoech (2009) noted that rESWT caused no pain, and neither local or generalized infections were observed throughout the observation period. Sixteen out of the 21 wounds healed within a mean period of six weeks (range: 3 to 9 weeks). In three cases, sufficient granulation tissue was formed after eight weeks on average, allowing for wound covering by gap tissue transplant. On average the size of the ulcers was reduced to 67% (20-100%) after the first week, 53% (15-90%) after the second week and 35% (9-78%) after the third week compared to baseline. These data indicate that the application of repetitive rESWT using the Swiss DolorClast is a low-effort and effective complement to standard therapy in diabetic foot ulcers without signs of infection or ischemia. In the study by Zoech (2009) patients were specifically very satisfied by the good tolerability and the absence of any significant side effects.

However, Zoech (2009) did not investigate a control group. Accordingly, it is currently unknown whether rESWT as performed by Zoech (2009) is more effective than sham-treatment of chronic soft tissue wounds. The present study was designed to answer this question.

ELIGIBILITY:
Inclusion Criteria:

* adults (both male and female) with chronic soft tissue wounds
* age range: between 18 and 80 years
* willingness of the patient to participate in the study, and written informed consent signed and personally dated by the patient
* different kinds of chronic soft tissue wounds: diabetic foot ulcers, post traumatic, venous stasis ulcer, decubitus
* wounds scored as Grade/Stage 1A, 1C, 2A and 2C according to Armstrong et al. (Diabetes Care 1998;21:855-859)
* No contraindications for rESWT

Exclusion Criteria:

* children and teenagers below the age of 18
* no willingness of the patient to participate in the study, and/or written informed consent not signed and not personally dated by the patient
* wounds scored as Grade/Stage 0A, 0B, 0C, 0D, 1B, 1D, 2B, 2D, 3A, 3B, 3C or 3D according to Armstrong et al. (1998)
* Burn wounds
* Uncontrolled diabetes because glycaemic control is crucial for wound healing and erratic values will effect the study results
* Blood sugar levels of the patient before meals are NOT regularly higher than 7mmol/L and are NOT regularly higher than 11mmol/L one to two hours after meals)
* Contraindications of rESWT: treatment of (i) soft tissue wounds over air-filled tissue (lung, gut), (ii) pregnant patients, (iii) patients with blood-clotting disorders (including local thrombosis), (iv) patients treated with oral anticoagulations, (v) soft tissue wounds above local tumors, and (vi) patients treated with local corticosteroid applications in the time period of six weeks before the first rESWT session (if applicable).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-02-23 (Actual); Primary Completion 2017-12-15 (Estimated); Study Completion 2017-12-15 (Estimated)

PRIMARY OUTCOMES:
Wound size | Three months after start of the treatments
  Individual time necessary to convert a chronic soft tissue wound from Grade/Stage 1A, 1C, 2A or 2C according to Armstrong et al. (Diabetes Care 1998;21:855-859) into Grade/Stage 0A or 0C according to Armstrong et al. (1998) (i.e., lesion completely epithelialized).

SECONDARY OUTCOMES:
Comfort during treatment | Immediately after each treatment session
  Individual patient's comfort during treatment will be assessed using a scale ranging from 0 (maximum discomfort) to 10 (maximum comfort).
Pain intensity during treatment | Immediately after each treatment session
  Individual patient's pain during treatment will be assessed using a scale ranging from 0 (no pain at all) to 10 (maximum, unbearable pain).
Satisfaction | Three months after start of the treatments
  Individual patient's satisfaction at three months after the start of the treatments will be assessed using a scale ranging from 0 (maximum dissatisfaction) to 10 (maximum satisfaction).

CONTACTS AND LOCATIONS:
Overall Officials: Harikrishna KR Nair, MD, Principal Investigator — Hospital Kuala Lumpur, Malaysia
Locations (1):
- Wound Care Unit, Dept. of Internal Medicine, Kuala Lumpur Hospital, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No